CLINICAL TRIAL: NCT04206241
Title: Assessing the Feasibility, Acceptability and Effects Of HIV Birth Testing In Maternity Settings In Zimbabwe
Status: Completed | Type: Observational
Sponsor: Elizabeth Glaser Pediatric AIDS Foundation (Other)
Collaborators: UNITAID (Other)
Responsible Party: Sponsor
Other Study IDs: EG0219
Record Dates: First submitted 2019-12-18; First posted 2019-12-20 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: HIV/AIDS; Infant Morbidity; Perinatal HIV Infection; HIV Infections
Keywords: HIV; POC; EID
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High-risk infants: Mother answered yes to any of the following questions on a risk-screening tool:
  * Mother diagnosed with HIV in labor and delivery?
  * Mother start ART after 32 weeks' gestation?
  * Maternal viral load above 1000 copies/ml in the 3rd trimester?
  * Mother seroconvert during pregnancy?
  * Was the mother not adhering to ART during pregnancy?
  Interventions: Diagnostic Test: Point of care early infant diagnosis (POC EID)
- Low-risk infants: Mothers did not answer affirmatively to any of the four screening questions
  Interventions: Diagnostic Test: Point of care early infant diagnosis (POC EID)

INTERVENTIONS:
Diagnostic Test: Point of care early infant diagnosis (POC EID) — HIV testing where the blood sample is processed at either the facility itself or a nearby site that is closer to the facility than a laboratory. With POC EID, blood samples do not have to travel to the laboratory for processing.
  Other Names: POC EID

SUMMARY:
This study aims to assess the feasibility and, acceptability and effects of implementing HIV testing at birth testing using point-of-care (POC) HIV nucleic acid testing (NAT) in maternity settings.

DETAILED DESCRIPTION:
This Unitaid-funded study aims to assess the feasibility and, acceptability and effects of implementing HIV testing at birth testing using point-of-care (POC) HIV nucleic acid testing (NAT) in maternity settings. Outcomes measures will include age at uptake of testing, turnaround time from testing to caregiver result receipt, HIV positivity rate, and timing of ART initiation for HIV-positive infants. This study will compare outcomes between HIV-exposed at high vs low risk of maternal HIV transmission. The study will also assess the impact of POC birth testing on retention in care and impact on subsequent testing at 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

HIV-exposed infants (HEI)

* All HEI who access maternity/post-natal services within 48 hours of life
* Tested for HIV at birth using the POC NAT platform
* Caregiver provides informed consent for participation

Caregivers

* Mother/caregiver of an HEI who was offered POC EID at birth
* Able to provide informed consent to participate in the study

Health workers

* All health workers working in maternity services in the study sites
* Provides informed consent to be interviewed

Key informants (laboratory managers and program leads/focal persons)

* Health managers working in the field of pediatric HIV services or PMTCT
* Provides informed consent to be interviewed

Exclusion Criteria:

HIV-exposed infants (HEI)

* HEI tested for HIV using conventional EID at project sites
* HEI whose caregivers refuse birth testing
* HEI where the clinician deems there is a contra-indication for sample collection for birth testing (e.g. severe hemophilia)

Caregivers

* Caregivers of HEI who cannot legally provide consent to participate in the study

Health workers

* Healthcare workers who do not make use of EID or results of EID

Key informants

* Key informants who cannot legally provide consent to participate in the study

Max Age: 48 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: * HIV-exposed infants newly born at the selected sites or presenting in study sites within 48 hours after birth
  * Health care workers and phlebotomists who are currently employed in study sites who are involved in providing POC EID services
  * Laboratory managers and program leads/focal persons at the Ministry of Health
  * Mothers/caregivers of HEI delivered or presenting in study sites within 48 hours after birth
Sampling Method: Non-Probability Sample
Enrollment: 278833 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of eligible HEI who present to pilot facilities who receive POC EID testing at birth | 18 months
  Number of eligible HEI who received POC EID divided by the total number of eligible HEI

SECONDARY OUTCOMES:
Proportion of tested HEI whose caregivers receive results of the POC EID birth testing | 18 months
  Number of HEI whose caregivers received results of the POC EID birth testing, divided by the number of HEI who received POC EID birth testing
Average number of days between sample collection of HEI and results received by caregiver | 18 months
  Date HEI sample collected minus date results received
Proportion of HEI tested at birth who are HIV positive | 18 months
  Number of HEI tested at birth who are HIV positive divided by the number of HEI tested at birth
Proportion of HIV-infected infants tested at birth who are started on ART within 2 weeks of the birth test | 18 months
  Number of HIV-infected infants tested at birth who are started on ART within 2 weeks of the birth test, divided by the number of HIV-infected infants tested at birth
Average number of days between sample collection of HEI and initiation on ART for infants testing HIV-positive | 18 months
  Date of sample collection of HEI minus date of date of ART initiation on ART for infants testing HIV-positive
Proportion of infants testing HIV negative at birth and who return for testing at 6-8 weeks | 18 months
  Number of infants testing HIV-negative at birth who return for testing at 6-8 weeks, divided by the number of infants who tested HIV-negative at birth
Proportion of infants who test HIV-positive at 6-8 weeks of those who test negative at birth | 18 months
  Number of infants who test HIV-positive at 6-8 weeks divided by those who tested HIV-negative at birth
The retention in care of positively-identified infants on birth testing for the first 3 and/or 6 months of life | 18 months
  Number of infants who tested HIV-positive at birth in care at 3 and/or 6 months of life, divided by the number who tested HIV-positive at birth
Proportion of HEI tested at birth who meet criteria for high risk of vertical transmission | 18 months
  Number of HEI tested at birth who meet the criteria for high risk of vertical transmission divided by the number who meet the criteria for high risk of vertical transmission
Proportion of high-risk infants according to the risk screening tool who test HIV-positive at birth | 18 months
  Number of high-risk infants according to the risk screening tool who test HIV-positive at birth, divided by the number of high-risk infants according to the risk screening tool
Proportion of low-risk infants according to the risk screening tool who test HIV-positive at birth | 18 months
  Number of low-risk infants according to the risk screening tool who test HIV-positive at birth, divided by the number of low-risk infants according the risk screening tool

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Mahomva, MBCHB, MPH, Principal Investigator — Elizabeth Glaser Pediatric AIDS Foundation - Zimbabwe
Locations (10):
- Zimbabwe (10):
  - Beitbridge District Hospital, Beitbridge
  - Bindura Provincial Hospital, Bindura
  - Chegutu District Hospital, Chegutu
  - Norton Hospital, Chegutu
  - Chiredzi District Hospital, Chiredzi
  - Gweru Provincial Hospital, Gweru
  - Victoria Falls District Hospital, Hwange
  - Kadoma District Hospital, Kadoma
  - Kwekwe General Hospital, Kwekwe
  - Masvingo Provincial Hospital, Masvingo